CLINICAL TRIAL: NCT07033676
Title: Study on the Correlation Between Serum miR-455-5p Level and Cardiac Structure and Function Parameters in Patients With Hypertensive Heart Disease
Brief Title: Serum miR-455-5p and Cardiac Structure and Function Parameters in Patients With Hypertensive Heart Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Cai Sidong, Assistant research fellow, The University of Hong Kong-Shenzhen Hospital
Other Study IDs: caisd@hku-szh.org; 82300446 (Other Grant/Funding Number: National Science Foundation of China); 2022A1515111093 (Other Grant/Funding Number: Guangdong Basic and Applied Basic Research Foundation); RCBS20231211090745071 (Other Grant/Funding Number: Shenzhen Science and Technology Program)
Record Dates: First submitted 2023-12-08; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Heart Disease
Keywords: miR-455-5p; hypertensive heart disease
MeSH Terms: conditions — Hypertension; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertensive heart disease (HHD) is the leading cause of mortality and morbidity worldwide. In 2017, the prevalence of HHD worldwide was 217.9 per 100,000 people, an increase of 7.4% over 1990, which has brought huge financial burden and social and economic losses to the world. Therefore, HHD is a major public health challenge worldwide. In our previous studies, we found that miR-455-5p, a microRNA, could functioned as an inducer to promote cardiac hypertrophy. Because cardiac hypertrophy was a common phenomenon in patients with HHD, so it is interesting to clarify whether miR-455-5p could be employed as a marker to indicate the function and/or structure of heart in the development of HHD. Thus, the purpose of this study was to collect blood samples of hypertensive patients, as well as analysis the correlation between serum miR-455-5p level and cardiac function. The research could help doctors better predict the course of hypertensive heart disease and provide more effective treatments for different patients.

DETAILED DESCRIPTION:
The purpose of this study was to collect blood samples of hypertensive patients, in order to clarify the correlation between serum miR-455-5p level and cardiac function. Generally, by using q-PCR assay, miR-455-5p level of each participants will be collected. Besides, SBP, DBP, LVPWd, LVIDd, IVSTd was detected by echocardiography and EF, FS, LVMi, RWT level was further calculated by LVIDd, LVPWd and IVSTd. Finally, the correlation of miR-455-5p level of HHD patients and LVPWd, LVIDd, IVSTd, EF, FS, LVMi, RWT, SBP, DBP was analysed.

ELIGIBILITY:
Inclusion Criteria:

* 1. age ≥18 years; 2. male or female; 3. systolic blood pressure ≥140mmHg or (and) diastolic blood pressure > 90mmHg; 4. history of hypertension>1year, NYHA grade I-IV

Exclusion Criteria:

* hypertensive heart diseases patients with other metabolic diseases or congenital diseases were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients with hypertensive heart disease admitted to Hong-Kong University, Shenzhen Hospital from January 1 to March 10 in 2021 were included in our study. Hypertensive heart disease was defined using the International Classification of Diseases, Ninth and Tenth Revision (ICD-10) codes. Diseases coded as I11.0 and I11.9 in ICD-10 were identified as hypertensive heart disease[1-2].
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum miR-455-5p level | the miR-455-5p level is collected at week 0, 6, 12 and 24.
  concentration of microRNA-455-5p in 100ml serum was determined by Elisa assay.
Measurement of LVPWd and LVPWs | the LVPWd and LVPWs are collected at week 0, 6, 12 and 24.
  left ventricular posterior wall thickness in diastole state and systole state are measured and recorded by echocardiography and its affiliated software.
Measurement of LVIDd and LVIDs | the LVIDd and LVIDs are collected at week 0, 6, 12 and 24.
  left ventricular internal diameter in diastole state and systole state are measured and recorded by echocardiography and its affiliated software.
Measurement of IVSTd and IVSTs | the IVSTd and IVSTs are collected at week 0, 6, 12 and 24.
  interventricular septum in diastole state and systole state are measured and recorded by echocardiography and its affiliated software.
Calculation of LVMi | the LVMi is calculated at week 0, 6, 12 and 24.
  left ventricular mass index was calculated based on the formula: LVMi=LVM/BSA; For LVM, LVM(g)=0.8*1.04*[(IVSTd+LVPWd+LVIDd)^3-LVIDd^3]+0.6; For BSA, BSA=[Body height (cm)*Body weight (kg)/3600]^0.5； Diagnosis of LVH: LVMi(Male)>115g/m2；LVMi(Female)>95g/m2
Measurement of LVEF | the EF is calculated at week 0, 6, 12 and 24.
  left ventricular ejection fraction are measured and recorded by echocardiography and its affiliated software.
  Generally, LVEF is range from 50% to 70% is regarded as normal. If LVEF less than 50%, the patient is suspected to suffered cardiac systolic dysfunction.
Measurement of FS | the FS is calculated at week 0, 6, 12 and 24.
  Fractional shortening are measured and recorded by echocardiography and its affiliated software.
  Generally, FS is range from 25% to 45% is regarded as normal. If FS less than 25%, the patient is suspected to suffered cardiac systolic dysfunction.
SBP | the SBP is collected at week 0, 6, 12 and 24.
  systolic blood pressure was measured by sphygmomanometer. For patients whose SBP is higher than 140mmHg, the patients is regarded as hypertension.
DBP | the DBP is collected at week 0, 6, 12 and 24.
  diastolic blood pressure was measured by sphygmomanometer. For patients whose DBP is higher than 90mmHg, the patients is regarded as hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Assistant research fellow, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (1):
- the University of Hongkong-Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided